CLINICAL TRIAL: NCT03145038
Title: Relative Bioavailability and Food Effect Study With Vericiguat to Characterize the Pediatric Formulation in Adult Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18581; 2016-005074-35 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Single oral dose of 20 x 0.5 mg vericiguat high-dose pediatric formulation, fed, American breakfast
  Interventions: Drug: Vericiguat(BAY1021189, high-dose pediatric-formulation)_fed
- Treatment B (Experimental): Single oral dose of 20 x 0.5 mg vericiguat high-dose pediatric formulation, fasted
  Interventions: Drug: Vericiguat(BAY1021189, high-dose pediatric-formulation)_fasted
- Treatment C (Experimental): Single oral dose of 25 x 0.1 mg vericiguat high-dose pediatric formulation, fed, American breakfast
  Interventions: Drug: Vericiguat(BAY1021189, low-dose pediatric-formulation)_fed
- Treatment D (Active Comparator): Single oral dose of 10 mg vericiguat intact IR tablet, adult formulation, fed, American breakfast
  Interventions: Drug: Vericiguat(BAY1021189,10 mg IR film-coated tablets,intact)_fed;American breakfast
- Treatment E (Experimental): Single oral dose of 10 mg vericiguat crushed IR tablet, adult formulation, fed, American breakfast
  Interventions: Drug: Vericiguat(BAY1021189,10 mg IR film-coated tablets,crushed)_fed;American breakfast
- Treatment F (Experimental): Single oral dose of 10 mg vericiguat intact IR tablet, adult formulation, fed, continental breakfast
  Interventions: Drug: Vericiguat(BAY1021189,10 mg IR film-coated tablets,intact)_fed;Continental breakfast

INTERVENTIONS:
Drug: Vericiguat(BAY1021189, high-dose pediatric-formulation)_fed — Vericiguat high-dose pediatric formulation (fed; American breakfast), 10 mg given as 20 x 0.5 mg mini tablets
  Arms: Treatment A
Drug: Vericiguat(BAY1021189, high-dose pediatric-formulation)_fasted — Vericiguat high-dose pediatric formulation (fasted),10 mg given as 20 x 0.5 mg mini tablets
  Arms: Treatment B
Drug: Vericiguat(BAY1021189, low-dose pediatric-formulation)_fed — Vericiguat low-dose pediatric-formulation (fed; American breakfast), 2.5 mg given as 25 x 0.1 mg mini tablets
  Arms: Treatment C
Drug: Vericiguat(BAY1021189,10 mg IR film-coated tablets,intact)_fed;American breakfast — 10 mg IR tablet, intact (fed; American breakfast)
  Arms: Treatment D
Drug: Vericiguat(BAY1021189,10 mg IR film-coated tablets,crushed)_fed;American breakfast — 10 mg IR tablet, crushed (fed; American breakfast)
  Arms: Treatment E
Drug: Vericiguat(BAY1021189,10 mg IR film-coated tablets,intact)_fed;Continental breakfast — 10 mg IR tablet, intact (fed; Continental breakfast)
  Arms: Treatment F

SUMMARY:
Vericiguat is intended to be used for the treatment of cardiovascular diseases, especially heart failure. Heart failure also occurs in children. Therefore, a study testing vericiguat in the treatment of heart failure in paediatric patients is planned under the paediatric investigational plan (PIP). In order to administer vericiguat to children, a vericiguat paediatric formulation is needed. This paediatric formulation is characterized in this study prior to its use in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at informed consent
* Race: white
* Body Mass Index (BMI): above or equal 18.0 and below or equal 29.9 kg / m²

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Febrile illness within 1 week prior to the first study drug administration
* History of postural syncopes
* A history of relevant diseases of vital organs, of the central nervous system or other organs
* A history of relevant smell and / or taste disorders
* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Medical disorder that would impair the subject's ability to complete the study in the opinion of the investigator.
* Known gastro-intestinal disorders (e.g. stomach ulcers, duodenal ulcers, gastrointestinal bleeding) or inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Vericiguat area under the plasma concentration vs. time curve divided by dose (AUC/D) | 0 - 72 hours
  AUC is the area under the curve (mathematically known as definite integral) in a plot of concentration of vericiguat after single dose administration in blood plasma against time (pre-dose until 72 hours after administration). AUC from time 0 to the last data point greater than lower limit of quantification divided by dose (AUC(0-tlast)/D) will be used as primary parameter if AUC cannot be calculated for all profiles, or mean AUC from the last data point to infinity [AUC(tlast-∞)] >20% of AUC. AUC will be analyzed by means of descriptive statistics.
Vericiguat maximum plasma concentration divided by dose (Cmax/D)) | 0 - 72 hours
  Cmax is the maximum observed vericiguat concentration in measured plasma after single dose administration (pre-dose until 72 hours after administration). Cmax/D is the maximum observed drug concentration in measured matrix after single dose administration divided by dose.Cmax will be analyzed by means of descriptive statistics

SECONDARY OUTCOMES:
Number of Adverse Events | pre-dose until 7 to 14 days after last administration of vericiguat
  As a secondary objective of this study the numbers of AEs will be used to assess safety and tolerability of vericiguat.
  In a clinical study, an AE is any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation subject after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Individual listings of AEs will be provided. The incidence of treatment-emergent AEs an drug-related AEs, respectively, will be summarized by treatment using MedDRA terms (highly specific standardised medical terminology).
Palatability of the oro-dispersible tablets and the crushed IR tablets assessed by questionnaire | up to 5 minutes after drug administration
  As a secondary objective of this study the taste and texture of pediatric formulation (palatability) (mini tablets) and of the crushed IR tablet will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical-Research-Services Mönchengladbach GmbH, Mönchengladbach, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/